CLINICAL TRIAL: NCT06540443
Title: A Pilot Feasibility Study of MPB-2043 Enhanced Magnetic Resonance Imaging (MRI) for Nodal Staging in Subjects With Head and Neck Squamous Cell Carcinomas
Brief Title: Pilot Study of MPB-2043 Enhanced MRI for Nodal Staging in Head and Neck Squamous Cell Carcinomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MegaPro Biomedical Co. Ltd. (Industry)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: IOP-CT-006
Record Dates: First submitted 2024-07-10; First posted 2024-08-06 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Lymph Node Metastasis
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Lymphatic Metastasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose cohort 1 (Experimental): pre- and post-enhanced MRI
  Interventions: Drug: MPB-2043 of 0.5 mg/kg
- Dose cohort 2 (Experimental): pre- and post-enhanced MRI
  Interventions: Drug: MPB-2043 of 1.0 mg/kg
- Dose cohort 3 (Experimental): pre- and post-enhanced MRI
  Interventions: Drug: MPB-2043 of 2.0 mg/kg
- Dose cohort 4 (Experimental): pre- and post-enhanced MRI
  Interventions: Drug: MPB-2043 of 3.0 mg/kg

INTERVENTIONS:
Drug: MPB-2043 of 0.5 mg/kg — Participants will undergo MRI scans without the administration of a contrast agent (unenhanced MRI) and IV-infused MPB-2043 for 1 hour.
  Other Names: MPB-2043 enhanced MRI
  Arms: Dose cohort 1
Drug: MPB-2043 of 1.0 mg/kg — Participants will undergo MRI scans without the administration of a contrast agent (unenhanced MRI) and IV-infused MPB-2043 for 1 hour.
  Other Names: MPB-2043 enhanced MRI
  Arms: Dose cohort 2
Drug: MPB-2043 of 2.0 mg/kg — Participants will undergo MRI scans without the administration of a contrast agent (unenhanced MRI) and IV-infused MPB-2043 for 1 hour.
  Other Names: MPB-2043 enhanced MRI
  Arms: Dose cohort 3
Drug: MPB-2043 of 3.0 mg/kg — Participants will undergo MRI scans without the administration of a contrast agent (unenhanced MRI) and IV-infused MPB-2043 for 1 hour.
  Other Names: MPB-2043 enhanced MRI
  Arms: Dose cohort 4

SUMMARY:
This study evaluates the safety and effectiveness of MPB-2043, a superparamagnetic iron oxide (SPIO) contrast agent, for enhancing MRI in detecting metastatic lymph nodes in head and neck cancer. The study compares four doses of MPB-2043 (0.5 mg/kg, 1 mg/kg, 2 mg/kg, and 3 mg/kg) and assesses the optimal timing for post-dose imaging using T1/T2/T2*-weighted sequences to improve the accuracy of nodal staging.

DETAILED DESCRIPTION:
The accurate detection of metastatic lymph nodes in subjects with head and neck squamous cell carcinomas is essential for appropriate staging and treatment planning. Traditional imaging techniques often struggle with detecting small nodal metastases due to limitations in resolution and contrast. Superparamagnetic iron oxide (SPIO) particles, such as MPB-2043, have shown promise as MRI contrast agents, particularly in the detection of metastatic lesions in the liver. This study extends the application of SPIO-enhanced MRI to the detection of metastatic cervical lymph nodes.

In this study, T1/T2/T2*-weighted MRI sequences will be used to assess signal intensity (SI) changes in lymph nodes after the administration of MPB-2043. The susceptibility effects of the iron oxide core cause tissue signal loss, which is more pronounced in normal lymph nodes taken up by the reticuloendothelial system, allowing for differentiation from malignant lymph nodes. The study will evaluate the safety and effectiveness of four different doses of MPB-2043 (0.5 mg/kg, 1 mg/kg, 2 mg/kg, and 3 mg/kg) in enhancing the visualization of cervical lymph nodes and will determine the most appropriate timing for post-dose imaging.

The primary objectives include determining the dose that provides optimal contrast enhancement without compromising safety and identifying the time points post-injection that offer the best differentiation between malignant and non-malignant lymph nodes. The results of this pilot feasibility study will inform the development of more extensive clinical trials aimed at improving the diagnostic accuracy of MRI in patients with head and neck squamous cell carcinomas.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 20 years and above
* Subjects with histologically proven head and neck squamous cell carcinomas or with suspicious metastatic lymph nodes (≥ pathological T-stage 1 and 2) without previous treatment by surgery
* Based on the site's clinical practice, subjects require lymphadenectomy treatment within 8 weeks.
* Subjects must be nonlactating.
* Subjects must be able to understand and be willing to sign a written informed consent document.
* Subjects must be able to comply with the study protocol.

Exclusion Criteria:

* Subjects with contraindications to MRI
* Subjects with a serious allergic history or known allergy to similar ingredients of the study contrast agent (i.e., Gd-based, SPIO particles, and iodinated contrast agents).
* Subjects obtained gadolinium-enhanced MRI ≤ 7 days before the enrollment.
* Subjects who participated in another imaging-related clinical trial 30 days prior to the study enrollment.
* Subjects with active systemic infections, active and clinically significant cardiac diseases, active gastrointestinal ulcers, or medical conditions that may significantly affect action, adequate absorption, and elimination of investigational contrast agent.
* Subjects with kidney disease or impairment.
* Subjects with liver or spleen disease or impairment based on other clinical imaging, such as CT or gadolinium contrast MRI, and clinical laboratory results.
* Subjects with active hepatitis B or hepatitis C infection.
* Subjects with bone marrow disorders or a history of a bone marrow transplant.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of MPB-2043 Enhanced MRI in Detecting Lymph Node Metastasis | Measured at pre-injection (Baseline) and 24 hours post-injection.
  1. Sensitivity is the proportion of true positive lymph nodes (those confirmed as metastatic by pathology) correctly identified by MPB-2043 enhanced MRI. A signal intensity change of 20% on T2*-weighted sequences post-injection is considered indicative of metastasis.
  2. Specificity is the proportion of true negative lymph nodes (those confirmed as non-metastatic by pathology) correctly identified by MPB-2043 enhanced MRI. A signal intensity change ≥ 50% on T2*-weighted sequences post-injection is considered indicative of non-metastasis.

SECONDARY OUTCOMES:
Changes in Signal Intensity of Lymph Nodes in Head and Neck MRI | From baseline to 10 minutes post-injection, and 24 hours post-injection.
  This outcome measure will assess and compare the changes in signal intensity (SI) in MRI images of lymph nodes in the head and neck region taken before and after the administration of MPB-2043.
  The SI changes will be evaluated across T1, T2, and T2*-weighted sequences.
Number and Size of Lymph Nodes Detected in Head and Neck | Measured at pre-injection (Baseline) and 24 hours post-injection.
  This outcome measure will record and evaluate the number and size of lymph nodes detected in the head and neck region/level via MRI post-administration of MPB-2043. The effectiveness of MPB-2043 in enhancing lymph node visibility and characterization will be determined by comparing these parameters before and after administration.
Determination of Optimal MPB-2043 Dosage for Lymph Node Imaging in Head and Neck MRI | Measured at pre-injection (Baseline) and 24 hours post-injection.
  This outcome measure will determine the most suitable dosage of MPB-2043 (0.5 mg/kg, 1 mg/kg, 2 mg/kg, 3 mg/kg) for optimal MRI contrast enhancement of lymph nodes in the head and neck region. The assessment will be based on post-dose MRI results, specifically evaluating signal intensity changes at 24 hours post-administration.
Safety Variables of Adverse Events | From baseline to Day 28 post-MPB-2043 administration.
  • The incidence of all adverse events
  * Treatment-emergent adverse events (AEs)
  * Serious AEs
  * Any AEs leading to withdrawal of study treatment
  * Any AEs leading to study discontinuation
  * Any AEs leading to death
  The data will be categorized and reported based on severity (mild, moderate, severe) and relatedness to the study drug, using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Safety Variables of Clinical Laboratory Tests | From baseline to Day 28 post-MPB-2043 administration.
  Clinical laboratory and vital sign data will be assessed for safety.
  This outcome measure evaluates the incidence of abnormal findings in clinical laboratory tests following the administration of MPB-2043. The tests include hematology (e.g., complete blood count), biochemistry (e.g., liver and kidney function tests), coagulation profiles (e.g., PT, INR, aPTT), and urinalysis. Results will be categorized as 'Normal,' 'Abnormal, Not Clinically Significant (NCS),' or 'Abnormal, Clinically Significant (CS).'

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jen Lou, MD., PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No